CLINICAL TRIAL: NCT07243210
Title: Effect of Irrigation Solution Temperature on Clinical Outcomes and Salivary CRP After Impacted Mandibular Third Molar Surgery: A Randomized Controlled Clinical Trial
Brief Title: Effect of Irrigation Solution Temperature on Clinical Outcomes and Salivary CRP After Impacted Mandibular Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Huynh Thien An, Lecturer, Department of Oral Surgery, Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Irrigation-CRP-2025; 269/2024/HĐ-ĐHYD (Other Grant/Funding Number: University of Medicine and Pharmacy at Ho Chi Minh City)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Third Molar Surgery; Postoperative Complications; C-REACTIVE PROTEIN
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Saline Irrigation (Experimental)
  Interventions: Procedure: Cold Saline Irrigation
- Room-Temperature Saline Irrigation (Active Comparator)
  Interventions: Procedure: Room-Temperature Saline Irrigation (Control)

INTERVENTIONS:
Procedure: Cold Saline Irrigation — During surgical extraction of impacted mandibular third molars, bone removal and irrigation will be performed using sterile saline cooled to 0-4°C to minimize heat generation
  Arms: Cold Saline Irrigation
Procedure: Room-Temperature Saline Irrigation (Control) — During surgical extraction of impacted mandibular third molars, bone removal and irrigation will be performed using sterile saline at room temperature (approximately 25°C). This procedure serves as the control to compare the effects of irrigation temperature on postoperative outcomes.
  Arms: Room-Temperature Saline Irrigation

SUMMARY:
Surgical extraction of impacted mandibular third molars often requires bone removal using rotary instruments, in which friction between the bur and bone generates heat. Excessive temperature rise may lead to local bone necrosis, delayed healing, and increased postoperative complications. Continuous irrigation with saline solution is routinely performed to reduce heat generation, and cold saline irrigation (0-4℃) has been shown to provide better thermal control than room-temperature saline.

This study aims to evaluate the effect of cold saline irrigation compared with room-temperature saline irrigation on postoperative outcomes following impacted mandibular third molar surgery. The assessed parameters include pain, swelling, trismus, and salivary C-reactive protein (CRP) levels as a biomarker of inflammation. Salivary CRP serves as a minimally invasive marker that reflects the systemic inflammatory response after surgery.

This randomized controlled trial will be conducted at the University of Medicine and Pharmacy at Ho Chi Minh City. Eligible patients with bilateral impacted mandibular third molars will be enrolled. Each patient will undergo extraction of one tooth with cold saline irrigation (0-4℃) and the contralateral tooth with room-temperature saline irrigation. Postoperative outcomes will include pain intensity (VAS) on days 1, 2, and 7; facial swelling on days 1, 2, and 7; trismus on days 1, 2, and 7; and salivary CRP levels at baseline and postoperative day 2.

The findings are expected to clarify the role of irrigation solution temperature in both subjective clinical outcomes and objective inflammatory markers, thereby providing evidence to optimize clinical protocols and reduce postoperative morbidity in third molar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with an ASA physical status classification of I or II.
* Patients with bilaterally impacted mandibular third molars of comparable difficulty, with an angulation difference between the two teeth not exceeding 15 degrees, confirmed by clinical and panoramic radiographic examination.
* Patients who have provided written informed consent after being fully informed about the study purpose and procedures.

Exclusion Criteria:

* Patients presenting with systemic or local acute inflammation or infection at the surgical site.
* Patients with systemic diseases contraindicating surgical tooth extraction.
* Patients with a history of corticosteroid or anti-inflammatory drug use within 3 weeks prior to participation.
* Patients with clinical or radiographic signs suggestive of tumors (benign or malignant) associated with or adjacent to the impacted mandibular third molar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Facial Swelling | Baseline (preoperative) and postoperative days 1, 2, and 7
  Facial swelling will be assessed by measuring three linear distances between standard facial landmarks: (1) tragus to pogonion, (2) gonion to lateral canthus, and (3) gonion to commissure.
  Postoperative swelling is measured as the change in facial dimension at each time point compared with the baseline measurement.
Postoperative Pain | Day 1, Day 2, and Day 7 after surgery
  Postoperative pain will be assessed using a 10-point Visual Analog Scale (VAS), where 0 represents no pain and 10 represents the worst imaginable pain.
Trismus | Baseline (preoperative) and postoperative days 1, 2, and 7
  Trismus will be evaluated by measuring the maximum interincisal distance (in millimeters) between the incisal edges of the upper and lower central incisors using a calibrated caliper.
  The degree of trismus will be determined by the reduction in mouth opening compared with the baseline (preoperative) measurement.
Salivary C-Reactive Protein (sCRP) Levels | Baseline and postoperative day 2
  Salivary C-reactive protein (sCRP) levels will be quantified using the ELISA method following the manufacturer's protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No